CLINICAL TRIAL: NCT02601365
Title: A Phase I Study of Inhaled GM-CSF in the Treatment of Respiratory Virus-associated Severe Pneumonia
Brief Title: Inhaled GM-CSF for Respiratory Virus-Associated Severe Pneumonia
Acronym: iGRASP
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Clinical Hold FDA
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSHCH0001
Record Dates: First submitted 2015-11-06; First posted 2015-11-10 (Estimated); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Acute Respiratory Distress Syndrome; Pneumonia; Respiratory Virus Infection
MeSH Terms: conditions — Respiratory Distress Syndrome; Pneumonia | interventions — sargramostim; KPNA1 protein, human

STUDY DESIGN:
Intervention Model Description: Phase I, open label dose escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aerosolized Sargramostim (Experimental): A self-controlled, open-label study to evaluate safety of Sargramostim administered by nebulization
  Interventions: Drug: Sargramostim 0.04 mcg/kg/dose; Drug: Sargramostim 0.2mcg/kg/dose; Drug: Sargramostim 1 mcg/kg/dose

INTERVENTIONS:
Drug: Sargramostim 0.04 mcg/kg/dose — The final dilution of sargramostim will occur at the bedside by a study team member. Cohort 1 will receive sargramostim 0.04 mcg/kg/dose nebulized to the inspiratory loop of the patients' mechanical ventilator circuit for 15 minutes.
  Other Names: Cohort 1
Drug: Sargramostim 0.2mcg/kg/dose — The final dilution of sargramostim will occur at the bedside by a study team member. Cohort 1 will receive sargramostim 0.2 mcg/kg/dose nebulized to the inspiratory loop of the patients' mechanical ventilator circuit for 15 minutes.
  Other Names: Cohort 2
Drug: Sargramostim 1 mcg/kg/dose — The final dilution of sargramostim will occur at the bedside by a study team member. Cohort 1 will receive sargramostim 1 mcg/kg/dose nebulized to the inspiratory loop of the patients' mechanical ventilator circuit for 15 minutes.
  Other Names: Cohort 3

SUMMARY:
This study will investigate the safety and efficacy of the administration of inhaled GM-CSF to patients with respiratory virus-associated pneumonia.

ELIGIBILITY:
Inclusion Criteria

Individuals must meet all of the following criteria to be eligible for inclusion in this study:

Male or female Age ≥ 18 years and ≤ 80 years Able to understand and willing to sign a written informed consent document, or if incapacitated, has a designated legal representative who is able to understand and willing to sign a written informed consent document Able and willing to adhere to study visit schedule and study procedures Currently either oro-tracheally or naso-tracheally intubated

Diagnosis of respiratory viral infection determined by:

Polymerase Chain Reaction (PCR)-based Respiratory Virus Panel (RVP) positive for at least one of the following:

Respiratory syncytial virus (RSV) Influenza A/B Parainfluenza 1/2/3 Human Metapneumovirus Adenovirus Rhinovirus

Exclusion criteria Individuals meeting any of the following criteria will be excluded from participating in this study.

Active tracheostomy History of either autoimmune PAP or primary genetic PAP diagnosis History of the presence of histopathologically- or radiographically-documented, clinically significant pulmonary fibrosis History of clinically significant cardiovascular disease including but not limited to Congestive heart failure associated with New York Heart Association (NYHA) Functional Classification of >1 (i.e., with any degree of symptoms) History of typical or atypical angina within the past 6 months regardless of possible relief by nitrates History of clinically significant coagulopathy, bleeding diathesis, or other hematological disease History of severe allergic or anaphylactic reaction to sargramostim, other yeast-derived products, or any component of the study drug History of any other serious medical condition that, in the opinion of the Principal Investigator, would interfere with the ability of the patient to complete the study Concomitant current or recent prior use of specific medications including Lithium, either active or prior use within two weeks of screening and/or enrollment Active non-steroidal anti-inflammatory drug use, including but not limited to ibuprofen Women who are pregnant (i.e. have a positive serum pregnancy test), intending to become pregnant, breast feeding, or women of child-bearing potential who are unwilling to use contraception or maintain abstinence during the course of the study History of active tobacco/marijuana/e-cigarette use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events of Inhaled Sargramostim in Adult Patients with Severe Respiratory Viral Pneumonia | 1 year
  The occurrence of any treatment-emergent Adverse Events (AE's) or Serious Adverse Events (SAE's) will be recorded over the course of the trial.

REFERENCES:
- [Background] Thomas NJ, Shaffer ML, Willson DF, Shih MC, Curley MA. Defining acute lung disease in children with the oxygenation saturation index. Pediatr Crit Care Med. 2010 Jan;11(1):12-7. doi: 10.1097/PCC.0b013e3181b0653d. PMID 19561556
- [Background] Cakarova L, Marsh LM, Wilhelm J, Mayer K, Grimminger F, Seeger W, Lohmeyer J, Herold S. Macrophage tumor necrosis factor-alpha induces epithelial expression of granulocyte-macrophage colony-stimulating factor: impact on alveolar epithelial repair. Am J Respir Crit Care Med. 2009 Sep 15;180(6):521-32. doi: 10.1164/rccm.200812-1837OC. Epub 2009 Jul 9. PMID 19590023
- [Background] Huang FF, Barnes PF, Feng Y, Donis R, Chroneos ZC, Idell S, Allen T, Perez DR, Whitsett JA, Dunussi-Joannopoulos K, Shams H. GM-CSF in the lung protects against lethal influenza infection. Am J Respir Crit Care Med. 2011 Jul 15;184(2):259-68. doi: 10.1164/rccm.201012-2036OC. Epub 2011 Apr 7. PMID 21474645
- [Background] Sever-Chroneos Z, Murthy A, Davis J, Florence JM, Kurdowska A, Krupa A, Tichelaar JW, White MR, Hartshorn KL, Kobzik L, Whitsett JA, Chroneos ZC. GM-CSF modulates pulmonary resistance to influenza A infection. Antiviral Res. 2011 Nov;92(2):319-28. doi: 10.1016/j.antiviral.2011.08.022. Epub 2011 Sep 8. PMID 21925209
- [Background] Ghoneim HE, Thomas PG, McCullers JA. Depletion of alveolar macrophages during influenza infection facilitates bacterial superinfections. J Immunol. 2013 Aug 1;191(3):1250-9. doi: 10.4049/jimmunol.1300014. Epub 2013 Jun 26. PMID 23804714
- [Background] Steinwede K, Tempelhof O, Bolte K, Maus R, Bohling J, Ueberberg B, Langer F, Christman JW, Paton JC, Ask K, Maharaj S, Kolb M, Gauldie J, Welte T, Maus UA. Local delivery of GM-CSF protects mice from lethal pneumococcal pneumonia. J Immunol. 2011 Nov 15;187(10):5346-56. doi: 10.4049/jimmunol.1101413. Epub 2011 Oct 14. PMID 22003204
- [Background] Unkel B, Hoegner K, Clausen BE, Lewe-Schlosser P, Bodner J, Gattenloehner S, Janssen H, Seeger W, Lohmeyer J, Herold S. Alveolar epithelial cells orchestrate DC function in murine viral pneumonia. J Clin Invest. 2012 Oct;122(10):3652-64. doi: 10.1172/JCI62139. Epub 2012 Sep 10. PMID 22996662
- [Background] Hall MW, Knatz NL, Vetterly C, Tomarello S, Wewers MD, Volk HD, Carcillo JA. Immunoparalysis and nosocomial infection in children with multiple organ dysfunction syndrome. Intensive Care Med. 2011 Mar;37(3):525-32. doi: 10.1007/s00134-010-2088-x. Epub 2010 Dec 10. PMID 21153402
- [Background] Paine R 3rd, Standiford TJ, Dechert RE, Moss M, Martin GS, Rosenberg AL, Thannickal VJ, Burnham EL, Brown MB, Hyzy RC. A randomized trial of recombinant human granulocyte-macrophage colony stimulating factor for patients with acute lung injury. Crit Care Med. 2012 Jan;40(1):90-7. doi: 10.1097/CCM.0b013e31822d7bf0. PMID 21926600
- [Background] Luisetti M, Kadija Z, Mariani F, Rodi G, Campo I, Trapnell BC. Therapy options in pulmonary alveolar proteinosis. Ther Adv Respir Dis. 2010 Aug;4(4):239-48. doi: 10.1177/1753465810378023. Epub 2010 Jul 20. PMID 20647242
- [Background] Trapnell BC, Carey BC, Uchida K, Suzuki T. Pulmonary alveolar proteinosis, a primary immunodeficiency of impaired GM-CSF stimulation of macrophages. Curr Opin Immunol. 2009 Oct;21(5):514-21. doi: 10.1016/j.coi.2009.09.004. Epub 2009 Sep 30. PMID 19796925
- [Background] Tazawa R, Trapnell BC, Inoue Y, Arai T, Takada T, Nasuhara Y, Hizawa N, Kasahara Y, Tatsumi K, Hojo M, Ishii H, Yokoba M, Tanaka N, Yamaguchi E, Eda R, Tsuchihashi Y, Morimoto K, Akira M, Terada M, Otsuka J, Ebina M, Kaneko C, Nukiwa T, Krischer JP, Akazawa K, Nakata K. Inhaled granulocyte/macrophage-colony stimulating factor as therapy for pulmonary alveolar proteinosis. Am J Respir Crit Care Med. 2010 Jun 15;181(12):1345-54. doi: 10.1164/rccm.200906-0978OC. Epub 2010 Feb 18. PMID 20167854
- [Background] Herold S, Hoegner K, Vadasz I, Gessler T, Wilhelm J, Mayer K, Morty RE, Walmrath HD, Seeger W, Lohmeyer J. Inhaled granulocyte/macrophage colony-stimulating factor as treatment of pneumonia-associated acute respiratory distress syndrome. Am J Respir Crit Care Med. 2014 Mar 1;189(5):609-11. doi: 10.1164/rccm.201311-2041LE. No abstract available. PMID 24579839
- [Background] Papiris SA, Tsirigotis P, Kolilekas L, Papadaki G, Papaioannou AI, Triantafillidou C, Papaporfyriou A, Karakatsani A, Kagouridis K, Griese M, Manali ED. Long-term inhaled granulocyte macrophage-colony-stimulating factor in autoimmune pulmonary alveolar proteinosis: effectiveness, safety, and lowest effective dose. Clin Drug Investig. 2014 Aug;34(8):553-64. doi: 10.1007/s40261-014-0208-z. PMID 24890235